CLINICAL TRIAL: NCT00446420
Title: Cognitive Impairment Following Sedation for Colonoscopy With Propofol, Midazolam and Fentanyl Combinations
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Melbourne Health (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 2006.228
Record Dates: First submitted 2007-03-08; First posted 2007-03-12 (Estimated); Last update posted 2013-05-30 (Estimated); Status verified 2013-05

CONDITIONS: Cognitive Impairment
MeSH Terms: conditions — Cognitive Dysfunction | interventions — Propofol; Midazolam; Fentanyl

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Active Comparator): These patients will only receive intravenous propofol which will be titrated to an OAA/S score of 3. They will not receive fentanyl, midazolam or any other drugs
  Interventions: Drug: Propofol, midazolam, fentanyl
- 2 (Active Comparator): These patients will receive propofol plus midazolam and/or fentanyl. Midazolam and fentanyl will be given in fixed doses first and propofol will be titrated to effect. All drugs will be given intravenously.
  Interventions: Drug: Propofol, midazolam, fentanyl

INTERVENTIONS:
Drug: Propofol, midazolam, fentanyl — All drugs administered in doses according to anaesthetists' discretion during sedation for colonoscopy
  Other Names: Diprivan; Sublimase; Versed

SUMMARY:
Our hypothesis is that adding midazolam and/or fentanyl to propofol sedation for elective outpatient colonoscopy increases cognitive impairment at hospital discharge without improving intraoperative conditions or reducing intraoperative side-effects.

200 healthy patients aged 18 years or older will be randomised to receive propofol or propofol plus midazolam and/or fentanyl. Cognitive impairment will be tested at hospital discharge using Cogstate computerised testing software.

DETAILED DESCRIPTION:
A great variety of drug combinations are administered to patients having elective outpatient colonoscopy. In addition, as patients are going home, some may have residual cognitive deficits that making leaving the hospital unsafe. This study aims to find drugs combinations that are associated with the least cognitive impairment.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 years or older presenting for elective outpatient colonoscopy following full bowel preparation

Exclusion Criteria:

* No cognitive impairment
* Adequate English language comprehension
* Not combined with other procedures

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2007-02; Primary Completion 2008-02 (Actual); Study Completion 2008-02 (Actual)

PRIMARY OUTCOMES:
Cognitive impairment at hospital discharge after elective outpatient colonoscopy | Before discharge from daycare facility

SECONDARY OUTCOMES:
Dreaming during sedation, intraoperative operating conditions and complications, satisfaction with care | Before discharge from daycare facility

CONTACTS AND LOCATIONS:
Overall Officials: Kate Leslie, MD, Principal Investigator — Melbourne Health
Locations (1):
- Royal Melbourne Hospital, Parkville, Victoria, Australia

REFERENCES:
- [Derived] Padmanabhan U, Leslie K, Eer AS, Maruff P, Silbert BS. Early cognitive impairment after sedation for colonoscopy: the effect of adding midazolam and/or fentanyl to propofol. Anesth Analg. 2009 Nov;109(5):1448-55. doi: 10.1213/ane.0b013e3181a6ad31. Epub 2009 Jul 17. PMID 19617584